CLINICAL TRIAL: NCT05581290
Title: AI-Flex: An Artificial Neural Network Integrated Flexible Multi-Modal Sensor Patch for Real-Time Continuous Physiological Monitoring and Inference
Brief Title: A Study of a Multi-Modal Sensor Patch for Real-Time Physiological Monitoring and Inference
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Imon Banerjee, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 22-005307
Record Dates: First submitted 2022-10-12; First posted 2022-10-14 (Actual); Last update posted 2024-05-23 (Actual); Status verified 2024-05

CONDITIONS: Cardiac Disease
Keywords: Underlying Cardiac Structural Condition
MeSH Terms: conditions — Heart Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Multi-Modal Sensor Patch Measurements (Experimental): Subjects referred to Mayo Clinic in Arizona Cardiology Clinic who have an underlying cardiac structural condition will have a 15-minute data collection via the prototype device, AI-Flex, and standard of care electrocardiogram (ECG), temperature, and photoplethysmogram (PPG) measurements.
  Interventions: Device: AI-Flex

INTERVENTIONS:
Device: AI-Flex — A flexible multi-modal bio-sensing device with integrated AI capability used to measure ECG (heart's electrical activity), body temperature, and PPG (blood volume in tissue); primarly mounted on the wrist and chest.

SUMMARY:
The purpose of this research is to validate the prototype AI-Flex device. Researchers at Mayo Clinic developed a new a flexible multi-modal bio-sensing device, AI-Flex, with integrated artificial intelligence (AI) capability. Integration of sensing and AI analysis on the same device removes the need for data storage on the cloud for later analysis. The goal of the device is to allow real-time monitoring of patient health and timely intervention based on patient health condition. It is hoped that the proposed flexible device will allow intimate skin contact using ultra-thin (<10 µm) geometry to reduce or eliminate relative movement between the skin and flexible epidermal sensors even during rapid motion of the subject, which would significantly improve the sensor signal quality for AI analysis.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be referred for Cardiology Clinic Visit.
* Subject must have underlying cardiac structural disease or condition to increase yield of clinically significant transmission
* Subject must be 18 - 85 years of age.

Exclusion Criteria:

- < 18 years of age or > 85 years of age.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2022-11-17 (Actual); Primary Completion 2023-11-17 (Actual); Study Completion 2023-11-17 (Actual)

PRIMARY OUTCOMES:
AI-Flex ECG Accuracy | Baseline
  Number of AI-Flex ECG interpretations to match the standard of care commercial ECG recording
AI-Flex Temperature Measurement Accuracy | Baseline
  Number of AI-Flex ECG interpretations to match the standard of care commercial temperature measurement
AI-Flex PPG Measurement Accuracy | Baseline
  Number of AI-Flex ECG interpretations to match the standard of care commercial photoplethysmogram (PPG) measurement

CONTACTS AND LOCATIONS:
Overall Officials: Imon Banerjee, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Imon Banerjee, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials